CLINICAL TRIAL: NCT03677947
Title: Inference-Based Cognitive Therapy Versus Exposure and Response Prevention for Obsessive-Compulsive Disorder: a 16-Session Randomized Controlled Trial
Brief Title: Inference-Based Cognitive Therapy Versus Exposure and Response Prevention for Obsessive-Compulsive Disorder
Acronym: RCT_TOC_16
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Frederick Aardema, Principal Investigator, Advanced Bionics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-1463
Record Dates: First submitted 2018-04-20; First posted 2018-09-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Obsessive-compulsive Disorders and Symptoms; Obsessive-Compulsive Disorder
Keywords: overvalued ideation; treatment acceptability; treatment adherence; treatment outcome; treatment resistance; treatment satisfaction; insight; cognitive therapy; inference based cognitive therapy; exposure and response prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: The RCT will compare the outcome of 16 sessions of IBCT compared to 16 sessions of ERP in OCD patients. The evaluators will be blind to the random allocation treatment conditions with a randomization ratio of 1:1. Both treatments will be administered by trained therapists on a weekly one-on-one basis over a 16-week period with 6-month follow-up conforming to current thinking on relapse in OCD. Conditions of treatment delivery, duration and monitoring will be equivalent across all groups. Both treatments are manualized and therapists will receive intensive training in one therapy protocol to ensure optimal delivery of each modality. Due to COVID-19, as of April, 2020, treatment will be delivered to participants by videoconferencing only. To protect the integrity and internal validity of the trial, participants who were recruited before this date and received the majority of treatment sessions in face-to-face physical meetings will be excluded from the principal statistical analyses.
Who Masked: Outcomes Assessor
Masking Description: The independent evaluators will be blind to the random allocation treatment conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inference-based cognitive therapy (Active Comparator): The treatment primarily targets the dysfunctional reasoning and overvalued ideas. IBCT does not include exposure, but aims to bring resolution to the initial obsessional doubt or overvalued idea by showing the participant that the obsession is the result of incorrect reasoning.
  Interventions: Other: Inference-based cognitive therapy
- Exposure and response prevention (Active Comparator): ERP is a treatment developed to help people confront their fears based on the rationale that exposure to feared objects, activities, or situations in a safe environment helps reduce fear and decrease avoidance. During the treatment, patients will engage in these exposures to feared stimuli within and between sessions according to hierarchies developed during the initial evaluation sessions, and refrain from engaging in compulsive behaviour until their anxiety subsides (i.e. ritual prevention).
  Interventions: Behavioral: Exposure and response prevention

INTERVENTIONS:
Behavioral: Exposure and response prevention — ERP is a treatment developed to help people confront their fears based on the rationale that exposure to feared objects, activities, or situations in a safe environment helps reduce fear and decrease avoidance. During the treatment, participants will engage in these exposures to feared stimuli within and between sessions according to hierarchies developed during the initial evaluation sessions, and refrain from engaging in compulsive behaviour until their anxiety subsides (i.e. ritual prevention). Exercises will consist of both exposure in vivo (i.e. exposure in real life situations) and/or imaginal exposure according to recommendations.
  Other Names: ERP
  Arms: Exposure and response prevention
Other: Inference-based cognitive therapy — The treatment primarily targets the dysfunctional reasoning that gives rise to obsessional doubts and overvalued ideas. IBCT does not include exposure in vivo, but instead, aims to bring resolution to the initial obsessional doubt or overvalued idea by showing the participant that the obsession is the result of incorrect reasoning.
  Other Names: IBCT
  Arms: Inference-based cognitive therapy

SUMMARY:
Obsessive-compulsive disorder (OCD) is a highly disabling psychiatric illness, characterized by obsessional thoughts that cause patients to perform time-consuming and distressing compulsive rituals. Exposure and Response Prevention (ERP) is a first-line psychological treatment of choice, which requires patients to face their fears by being exposed to feared stimuli. ERP has been shown to reduce symptoms among those who comply with treatment. However, there is still a significant portion of patients that do not improve, especially those who firmly believe their obsessions are realistic and reasonable (i.e. OCD with Overvalued Ideation (OVI)). Also, a signficant proportion of patients refuse the treatment or drop out during treatment due to the distress provoked by ERP. Even among those that do improve, residual symptoms often remain, or symptoms may reappear after treatment. One evidence-based approach to the treatment of OCD, termed inference-based cognitive therapy (IBCT) has been shown to be as effective as ERP with the potential to overcome some of the limitations of ERP. Since IBCT is a cognitive approach, the treatment does not require exposure to feared stimuli and likely more tolerable for patients with OCD. Also, there is evidence that IBCT is more effective than ERP for those with overvalued ideation, since it directly targets the distorted reasoning that is responsible for the intensity and persistence of the obsession. The current study aims to directly compare ERP with this promising evidence-based cognitive therapy, which is expected to be significantly more effective for those with overvalued ideation, as well as significantly more tolerable with lower rates of treatment refusal, drop-out and higher treatment satisfaction. The project is designed to maximize potential beneficial health outcomes and offer a new evidence-based treatment option for the large proportion of patients unable to benefit from ERP.

DETAILED DESCRIPTION:
The proposed study is a parallel-group randomized controlled trial developed in accordance with CONSORT quality guidelines.The RCT will compare the outcome of 16 sessions of IBCT compared to 16 sessions of ERP in OCD patients. The principal investigators and independent evaluators will be blind to the random allocation treatment conditions with a randomization ratio of 1:1. Both treatments will be administered by trained therapists on a weekly one-on-one basis over a 16-week period with 6-month follow-up conforming to current thinking on relapse in OCD. Conditions of treatment delivery, duration and monitoring will be equivalent across all groups. Both treatments are manualized and any newly engaged therapists will receive intensive training in one therapy protocol to ensure optimal delivery of each modality.

The objective of the present study is to establish IBCT as a psychological treatment that is as effective as ERP, but significantly more tolerable and generalizable for the high proportion of patients who are unable to benefit from ERP.

The hypotheses are that 1) IBCT is non-inferior to ERP; 2) IBCT is superior to ERP among OCD patients with higher levels of OVI; 3) IBCT has lower rates of treatment refusal and drop-out than ERP; and, 4) IBCT has higher levels of acceptability, tolerability, credibility and satisfaction than ERP.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of OCD according to Diagnostical and Statistical Manual, version 5 criteria;
* no change in medication during the 12 weeks before treatment for antidepressants (4 weeks for anxiolytics);
* willingness to keep medication stable while participating in the study;
* no evidence of suicidal intent;
* no evidence of current substance abuse;
* no evidence of current or past schizophrenia, bipolar disorder or organic mental disorder;
* not undergoing a current psychological treatment;
* willingness to undergo active psychological treatment;
* willingness to undergo randomization into treatment modality;
* fluency in English and French.

Exclusion criteria:

* another primary diagnosis than OCD requiring treatment;
* medication not stabilized for 12 weeks;
* medication will change during the participation;
* suicidal intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
assessment of change in obsessive and compulsive symptoms and severity | baseline measure of obsessive and compulsive symptoms of OCD
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a 10-item scale designed to measure the severity and type of symptoms in people with obsessive-compulsive disorder (OCD) over the past seven days. The symptoms assessed are obsessions and compulsions. This scale is useful in tracking OCD symptoms at intake and during/after treatment.
  Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms. Scores on the obsession and compulsion subscales range from 0 to 20, but only the total Y-BOCS score is interpreted. Total scores can be split into five categories, based on severity of symptoms. People who have a total Y-BOCS score:
  Under 7 are likely to be subclinical, 8-15 are likely to have a mild case of OCD, 16-23 are likely to have a moderate case of OCD, 24-31 are likely to have a severe case of OCD, 32-40 are likely to have an extreme case of OCD.
assessment of change in obsessive and compulsive symptoms and severity | up to 8 weeks
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a 10-item scale designed to measure the severity and type of symptoms in people with obsessive-compulsive disorder (OCD) over the past seven days. The symptoms assessed are obsessions and compulsions. This scale is useful in tracking OCD symptoms at intake and during/after treatment.
  Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms. Scores on the obsession and compulsion subscales range from 0 to 20, but only the total Y-BOCS score is interpreted. Total scores can be split into five categories, based on severity of symptoms. People who have a total Y-BOCS score:
  Under 7 are likely to be subclinical, 8-15 are likely to have a mild case of OCD, 16-23 are likely to have a moderate case of OCD, 24-31 are likely to have a severe case of OCD, 32-40 are likely to have an extreme case of OCD.
assessment of change in obsessive and compulsive symptoms and severity | up to 16 weeks
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a 10-item scale designed to measure the severity and type of symptoms in people with obsessive-compulsive disorder (OCD) over the past seven days. The symptoms assessed are obsessions and compulsions. This scale is useful in tracking OCD symptoms at intake and during/after treatment.
  Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms. Scores on the obsession and compulsion subscales range from 0 to 20, but only the total Y-BOCS score is interpreted. Total scores can be split into five categories, based on severity of symptoms. People who have a total Y-BOCS score:
  Under 7 are likely to be subclinical, 8-15 are likely to have a mild case of OCD, 16-23 are likely to have a moderate case of OCD, 24-31 are likely to have a severe case of OCD, 32-40 are likely to have an extreme case of OCD.
assessment of change in obsessive and compulsive symptoms and severity | change from baseline at 6 months
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a 10-item scale designed to measure the severity and type of symptoms in people with obsessive-compulsive disorder (OCD) over the past seven days. The symptoms assessed are obsessions and compulsions. This scale is useful in tracking OCD symptoms at intake and during/after treatment.
  Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms. Scores on the obsession and compulsion subscales range from 0 to 20, but only the total Y-BOCS score is interpreted. Total scores can be split into five categories, based on severity of symptoms. People who have a total Y-BOCS score:
  Under 7 are likely to be subclinical, 8-15 are likely to have a mild case of OCD, 16-23 are likely to have a moderate case of OCD, 24-31 are likely to have a severe case of OCD, 32-40 are likely to have an extreme case of OCD.
establishing baseline level of overvalued ideation | baseline measure
  The Over-Valued Ideas Scale (OVIS) is an 11-item clinician administered scale assess severity of overvalued ideation. These include how strong obsessive belief; how reasonable the belief is; how weak and strong the belief has fluctuated over the past week; how accurate the belief is; the extent to which others share the same beliefs; how the patient attributes similar or differing beliefs in other people; how effective and important the compulsions are; the extent to which their disorder has caused their obsessive belief; and their degree of resistance toward the belief on a 1 to 10 scale. The average of the 11 items provides an estimate of one's degree of OVI, where higher scores represent greater levels of OVI.
assess change in level of overvalued ideation | change from baseline at 8 weeks
  The Over-Valued Ideas Scale (OVIS) is an 11-item clinician administered scale assess severity of overvalued ideation. These include how strong obsessive belief; how reasonable the belief is; how weak and strong the belief has fluctuated over the past week; how accurate the belief is; the extent to which others share the same beliefs; how the patient attributes similar or differing beliefs in other people; how effective and important the compulsions are; the extent to which their disorder has caused their obsessive belief; and their degree of resistance toward the belief on a 1 to 10 scale. The average of the 11 items provides an estimate of one's degree of OVI, where higher scores represent greater levels of OVI.
assess change in level of overvalued ideation | change from baseline at 16 weeks
  The Over-Valued Ideas Scale (OVIS) is an 11-item clinician administered scale assess severity of overvalued ideation. These include how strong obsessive belief; how reasonable the belief is; how weak and strong the belief has fluctuated over the past week; how accurate the belief is; the extent to which others share the same beliefs; how the patient attributes similar or differing beliefs in other people; how effective and important the compulsions are; the extent to which their disorder has caused their obsessive belief; and their degree of resistance toward the belief on a 1 to 10 scale. The average of the 11 items provides an estimate of one's degree of OVI, where higher scores represent greater levels of OVI.
assess change in level of overvalued ideation | change from baseline at 6 months
  The Over-Valued Ideas Scale (OVIS) is an 11-item clinician administered scale assess severity of overvalued ideation. These include how strong obsessive belief; how reasonable the belief is; how weak and strong the belief has fluctuated over the past week; how accurate the belief is; the extent to which others share the same beliefs; how the patient attributes similar or differing beliefs in other people; how effective and important the compulsions are; the extent to which their disorder has caused their obsessive belief; and their degree of resistance toward the belief on a 1 to 10 scale. The average of the 11 items provides an estimate of one's degree of OVI, where higher scores represent greater levels of OVI.

OTHER OUTCOMES:
assessing change in symptoms of obsessive-compulsive disorder and associated personality | baseline measure
  The Vancouver Obsessional-Compulsive Inventory (VOCI) is a 55-item self-report measure designed to assess a broad spectrum of OCD symptoms and associated personality characteristics. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much), and measure participants' agreement with a series of statements related to obsessions and compulsions (e.g., ''I am often very upset by my unwanted impulses to harm other people''). The VOCI has six component subscales: (a) Checking; (b) Contamination; (c) Obsessions; (d) Hoarding; (e) ''Just Right''; and (f) Indecisiveness.
assessing change in symptoms of obsessive-compulsive disorder and associated personality | change from baseline at 8 weeks
  The Vancouver Obsessional-Compulsive Inventory (VOCI) is a 55-item self-report measure designed to assess a broad spectrum of OCD symptoms and associated personality characteristics. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much), and measure participants' agreement with a series of statements related to obsessions and compulsions (e.g., ''I am often very upset by my unwanted impulses to harm other people''). The VOCI has six component subscales: (a) Checking; (b) Contamination; (c) Obsessions; (d) Hoarding; (e) ''Just Right''; and (f) Indecisiveness.
assessing change in symptoms of obsessive-compulsive disorder and associated personality | change from baseline at 16 weeks
  The Vancouver Obsessional-Compulsive Inventory (VOCI) is a 55-item self-report measure designed to assess a broad spectrum of OCD symptoms and associated personality characteristics. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much), and measure participants' agreement with a series of statements related to obsessions and compulsions (e.g., ''I am often very upset by my unwanted impulses to harm other people''). The VOCI has six component subscales: (a) Checking; (b) Contamination; (c) Obsessions; (d) Hoarding; (e) ''Just Right''; and (f) Indecisiveness.
assessing change in symptoms of obsessive-compulsive disorder and associated personality | change from baseline at 6 months
  The Vancouver Obsessional-Compulsive Inventory (VOCI) is a 55-item self-report measure designed to assess a broad spectrum of OCD symptoms and associated personality characteristics. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much), and measure participants' agreement with a series of statements related to obsessions and compulsions (e.g., ''I am often very upset by my unwanted impulses to harm other people''). The VOCI has six component subscales: (a) Checking; (b) Contamination; (c) Obsessions; (d) Hoarding; (e) ''Just Right''; and (f) Indecisiveness.
assess change in symptoms of depression | baseline diagnosis to provide description of depression symptoms
  The Beck Depression Inventory, version II consists of 21 items assessing symptoms of depression experienced during the past 2 weeks. Each item contains four statements reflecting varying degrees of symptom severity. Respondents are instructed to circle the number (ranging from zero to three, indicating increasing severity) that corresponds with the statement that best describes them. Ratings are summed to calculate a total Beck Depression Inventory, version II score, which can range from 0 to 63.
assess change in symptoms of depression | change from baseline diagnosis to provide description of depression symptoms at the beginning of the treatment
  The Beck Depression Inventory, version II consists of 21 items assessing symptoms of depression experienced during the past 2 weeks. Each item contains four statements reflecting varying degrees of symptom severity. Respondents are instructed to circle the number (ranging from zero to three, indicating increasing severity) that corresponds with the statement that best describes them. Ratings are summed to calculate a total Beck Depression Inventory, version II score, which can range from 0 to 63.
assess change in symptoms of depression | change from beginning of the treatment at 8 weeks
  The Beck Depression Inventory, version II consists of 21 items assessing symptoms of depression experienced during the past 2 weeks. Each item contains four statements reflecting varying degrees of symptom severity. Respondents are instructed to circle the number (ranging from zero to three, indicating increasing severity) that corresponds with the statement that best describes them. Ratings are summed to calculate a total Beck Depression Inventory, version II score, which can range from 0 to 63.
assess change in symptoms of depression | change from beginning of the treatment at 16 weeks
  The Beck Depression Inventory, version II consists of 21 items assessing symptoms of depression experienced during the past 2 weeks. Each item contains four statements reflecting varying degrees of symptom severity. Respondents are instructed to circle the number (ranging from zero to three, indicating increasing severity) that corresponds with the statement that best describes them. Ratings are summed to calculate a total Beck Depression Inventory, version II score, which can range from 0 to 63.
assess change in symptoms of depression | change from beginning of the treatment at 6 months
  The Beck Depression Inventory, version II consists of 21 items assessing symptoms of depression experienced during the past 2 weeks. Each item contains four statements reflecting varying degrees of symptom severity. Respondents are instructed to circle the number (ranging from zero to three, indicating increasing severity) that corresponds with the statement that best describes them. Ratings are summed to calculate a total Beck Depression Inventory, version II score, which can range from 0 to 63.
assess change in symptoms of anxiety | baseline measure
  The Beck Anxiety inventory is a scale of 21 items describe the most typical symptoms of anxiety disorders. It was developed to measure the intensity of anxiety symptoms in clinical populations. It asks respondents to indicate how much they have been affected by each symptom during the last week, on a scale from 0 (Not at all) to 3 (Severely - I could barely stand it). Total scores are the sum of all item scores, and range from 0 to 63; higher scores indicate higher anxiety.
assess change in symptoms of anxiety | change from baseline at 8 weeks
  The Beck Anxiety inventory is a scale of 21 items describe the most typical symptoms of anxiety disorders. It was developed to measure the intensity of anxiety symptoms in clinical populations. It asks respondents to indicate how much they have been affected by each symptom during the last week, on a scale from 0 (Not at all) to 3 (Severely - I could barely stand it). Total scores are the sum of all item scores, and range from 0 to 63; higher scores indicate higher anxiety.
assess change in symptoms of anxiety | change from baseline at 16 weeks
  The Beck Anxiety inventory is a scale of 21 items describe the most typical symptoms of anxiety disorders. It was developed to measure the intensity of anxiety symptoms in clinical populations. It asks respondents to indicate how much they have been affected by each symptom during the last week, on a scale from 0 (Not at all) to 3 (Severely - I could barely stand it). Total scores are the sum of all item scores, and range from 0 to 63; higher scores indicate higher anxiety.
assess change in symptoms of anxiety | change from baseline at 6 months
  The Beck Anxiety inventory is a scale of 21 items describe the most typical symptoms of anxiety disorders. It was developed to measure the intensity of anxiety symptoms in clinical populations. It asks respondents to indicate how much they have been affected by each symptom during the last week, on a scale from 0 (Not at all) to 3 (Severely - I could barely stand it). Total scores are the sum of all item scores, and range from 0 to 63; higher scores indicate higher anxiety.
assess impairment in different domain | baseline measure
  The Sheehan Disability Scale is a standard measure of impairment in work, social life and family responsibilities which was a composite of 3 self-rated 10-point (0=none, l-3=mild, 4-6=moderate, 7-9=marked, and 10=extreme) Likert response items to assess work, family, and social functioning during the last month.
assess change in impairment in different domain | change from baseline at 16 weeks
  The Sheehan Disability Scale is a standard measure of impairment in work, social life and family responsibilities which was a composite of 3 self-rated 10-point (0=none, l-3=mild, 4-6=moderate, 7-9=marked, and 10=extreme) Likert response items to assess work, family, and social functioning during the last month.
assess change in impairment in different domain | change from baseline at 6 months
  The Sheehan Disability Scale is a standard measure of impairment in work, social life and family responsibilities which was a composite of 3 self-rated 10-point (0=none, l-3=mild, 4-6=moderate, 7-9=marked, and 10=extreme) Likert response items to assess work, family, and social functioning during the last month.
measure of health-related quality of life | baseline measure
  EuroQol-5dimensions is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5Dimensions consists of a descriptive system and the EQ Value Average Score.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ Value Average Score used as a quantitative measure of health outcome that reflects the participant's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
  The final score is a scale numbered from 0 to 100, where100 means the best health you can imagine and 0 means the worst health you can imagine.
measure of health-related quality of life | change from baseline at 16 weeks
  EuroQol-5dimensions is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5Dimensions consists of a descriptive system and the EQ Value Average Score.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ Value Average Score records the participant's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the participant's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
  The final score is a scale numbered from 0 to 100, where100 means the best health you can imagine and 0 means the worst health you can imagine.
measure of health-related quality of life | change from baseline at 6 months
  EuroQol-5dimensions is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5Dimensions consists of a descriptive system and the EQ Value Average Score.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EuroQuol Value Average Score records the participant's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the participant's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
  The final score is a scale numbered from 0 to 100, where100 means the best health you can imagine and 0 means the worst health you can imagine.
assessment of change in inferential confusion due to obsessive-compulsive disorder | baseline measure
  The Inferential Confusion Questionnaire-Expanded Version (ICQ-EV) is a 30-item questionnaire measuring an overreliance on imagination, a distrust of the senses, and a tendency to confuse imagination with reality during reasoning. Like the original version, the expanded version of the ICQ is a highly reliable measure that has been shown to explain a large portion of the variance in symptoms of OCD independent of negative mood states and other cognitive domains. Items are rated on a 6-point scale .
assessment of change in inferential confusion due to obsessive-compulsive disorder | change from baseline measure at 16 weeks
  The Inferential Confusion Questionnaire-Expanded Version (ICQ-EV) is a 30-item questionnaire measuring an overreliance on imagination, a distrust of the senses, and a tendency to confuse imagination with reality during reasoning. Like the original version, the expanded version of the ICQ is a highly reliable measure that has been shown to explain a large portion of the variance in symptoms of OCD independent of negative mood states and other cognitive domains. Items are rated on a 6-point scale .
assessment of change in inferential confusion due to symptoms of obsessive-compulsive disorder | change from baseline measure at 6 months
  The Inferential Confusion Questionnaire-Expanded Version (ICQ-EV) is a 30-item questionnaire measuring an overreliance on imagination, a distrust of the senses, and a tendency to confuse imagination with reality during reasoning. Like the original version, the expanded version of the ICQ is a highly reliable measure that has been shown to explain a large portion of the variance in symptoms of OCD independent of negative mood states and other cognitive domains. Items are rated on a 6-point scale .
measure change of obsessive beliefs | baseline measure
  The obsessive beliefs questionnaire is a 20-item key self report questionnaire measuring change in obsessive beliefs domains. Items are answered on a 7-point Likert-type scale (disagree very much to agree very much) in relation to "what you are like most of the time."
measure change of obsessive beliefs | change from baseline measure at 16 weeks
  The obsessive beliefs questionnaire is a 20-item key self report questionnaire measuring change in obsessive beliefs domains. Items are answered on a 7-point Likert-type scale (disagree very much to agree very much) in relation to "what you are like most of the time."
measure change of obsessive beliefs | change from baseline measure at 6 months
  The obsessive beliefs questionnaire is a 20-item key self report questionnaire measuring change in obsessive beliefs domains. Items are answered on a 7-point Likert-type scale (disagree very much to agree very much) in relation to "what you are like most of the time."
used to assess change in acceptability and adherence of treatment | baseline measure
  The Treatment Acceptability/Adherence Scale (TAAS) will be tested by comparing our indices of tolerability across the two treatments. It is a 10-item scale rated on a 7-point scale and assesses acceptability of and anticipated adherence to a given treatment. Higher scores represent greater acceptability.
used to assess change in acceptability and adherence of treatment | after 8 treatment session
  The Treatment Acceptability/Adherence Scale (TAAS) will be tested by comparing our indices of tolerability across the two treatments. It is a 10-item scale rated on a 7-point scale and assesses acceptability of and anticipated adherence to a given treatment. Higher scores represent greater acceptability.
used to assess change in acceptability and adherence of treatment | after 16 treatment session
  The Treatment Acceptability/Adherence Scale (TAAS) will be tested by comparing our indices of tolerability across the two treatments. It is a 10-item scale rated on a 7-point scale and assesses acceptability of and anticipated adherence to a given treatment. Higher scores represent greater acceptability.
used to evaluate credibility and expectancy of treatment modality by participant | baseline measure
  The Credibility and Expectancy Questionnaire (CEQ) is a 6-item measure divided into two subscales assessing treatment credibility (CEQ-Credibility) and expectancy (CEQ-Expectancy), respectively. The first three CEQ items assess credibility and are rated from 1 to 9 with total possible scores ranging from 3 to 27, where higher scores indicate greater credibility beliefs. The final three CEQ items assess expectancy, with one item rated from 1 to 9, and two items rated from 0% to 100% (values from 1 to 11). We standardized these three items into z scores before summing to create the total Expectancy score. The Expectancy scale scores ranged from -6.72 to 5.51, where higher scores indicate higher expectations.
used to evaluate credibility and expectancy of treatment modality by participant | up to 8 weeks
  The Credibility and Expectancy Questionnaire (CEQ) is a 6-item measure divided into two subscales assessing treatment credibility (CEQ-Credibility) and expectancy (CEQ-Expectancy), respectively. The first three CEQ items assess credibility and are rated from 1 to 9 with total possible scores ranging from 3 to 27, where higher scores indicate greater credibility beliefs. The final three CEQ items assess expectancy, with one item rated from 1 to 9, and two items rated from 0% to 100% (values from 1 to 11). We standardized these three items into z scores before summing to create the total Expectancy score. The Expectancy scale scores ranged from -6.72 to 5.51, where higher scores indicate higher expectations.
used to evaluate credibility and expectancy of treatment modality by participant | up to 16 weeks
  The Credibility and Expectancy Questionnaire (CEQ) is a 6-item measure divided into two subscales assessing treatment credibility (CEQ-Credibility) and expectancy (CEQ-Expectancy), respectively. The first three CEQ items assess credibility and are rated from 1 to 9 with total possible scores ranging from 3 to 27, where higher scores indicate greater credibility beliefs. The final three CEQ items assess expectancy, with one item rated from 1 to 9, and two items rated from 0% to 100% (values from 1 to 11). We standardized these three items into z scores before summing to create the total Expectancy score. The Expectancy scale scores ranged from -6.72 to 5.51, where higher scores indicate higher expectations.
used to evaluate the treatment satisfaction of the participant | baseline measure
  The Evaluation of Treatment Questionnaire is a 19-item subjective measure assessing treatment satisfaction. It is a qualitative and quantitative questionnaire. The first two items assess how far therapy help, their importance and the satisfaction. The second part rate what the participant think about the therapy in a 1 to 10 scale. The third part assess what participant feel about the therapy on different scale. Finally, the last part rate satisfaction, preoccupation, stress and what the less like about the therapy.
used to evaluate the treatment satisfaction of the participant | up to 8 weeks
  The Evaluation of Treatment Questionnaire is a 19-item subjective measure assessing treatment satisfaction. It is a qualitative and quantitative questionnaire. The first two items assess how far therapy help, their importance and the satisfaction of the participant. The second part rate what the participant think about the therapy in a 1 to 10 scale. The third part assess what participant feel about the therapy on different scale. Finally, the last part rate satisfaction, preoccupation, stress and what the participant less like about the therapy.
used to evaluate the treatment satisfaction of the participant | up to 16 weeks
  The Evaluation of Treatment Questionnaire is a 19-item subjective measure assessing treatment satisfaction. It is a qualitative and quantitative questionnaire. The first two items assess how far therapy help, their importance and the satisfaction. The second part rate what the participant think about the therapy in a 1 to 10 scale. The third part assess what participant feel about the therapy on different scale. Finally, the last part rate satisfaction, preoccupation, stress and what the less like about the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Aardema, Ph. D., Principal Investigator — Université de Montréal
Locations (1):
- Centre de recherche de l'Institut universitaire en santé mentale de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No